CLINICAL TRIAL: NCT04821154
Title: Clinical Investigation to Demonstrate Performance, Safety and Clinical Benefits of the Persona Revision Knee System
Brief Title: Persona Revision Knee System Outcomes
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMG2019-13K
Record Dates: First submitted 2021-03-23; First posted 2021-03-29 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2024-12

CONDITIONS: Arthroplasty Complications; Infection; Knee Disease; Knee Osteoarthritis
Keywords: Revision; Total Knee; Medical Device; Safety; Performance; Primary; Clinical Benefits
MeSH Terms: conditions — Infections; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (11):
- 1) Revision Splined CCK: Patients who were implanted with a splined tibial stem, 0 degree Persona Revision tibial component, constrained condylar knee (CCK) articular surface, Persona Revision femoral component, and splined femoral stem.
  Interventions: Device: Persona Revision Knee System
- 2) Revision Cemented CCK: Patients who were implanted with a cemented tibial stem, 0 degree Persona Revision tibial component, CCK articular surface, Persona Revision femoral component, and cemented femoral stem.
  Interventions: Device: Persona Revision Knee System
- 3) Revision Splined PS/CPS: Patients who were implanted with a splined tibial stem, 0 degree Persona Revision tibial component, posterior stabilized/constrained posterior stabilized (PS/CPS) articular surface, Persona Revision femoral component, and splined femoral stem.
  Interventions: Device: Persona Revision Knee System
- 4) Revision Cemented PS/CPS: Patients who were implanted with a cemented tibial stem, 0 degree Persona Revision tibial component, PS/CPS articular surface, Persona Revision femoral component, and cemented femoral stem.
  Interventions: Device: Persona Revision Knee System
- 5) Revision Splined PS/CPS: Patients who were implanted with a splined tibial stem, 0 degree Persona Revision tibial component, PS/CPS articular surface, Persona primary PS femoral component, with no femoral stem.
  Interventions: Device: Persona Revision Knee System
- 6) Revision Cemented PS/CPS: Patients who were implanted with a cemented tibial stem, 0 degree Persona Revision tibial component, PS/CPS articular surface, Persona primary PS femoral component, with no femoral stem.
  Interventions: Device: Persona Revision Knee System
- 7) Revision Cemented CCK with 5 Degree Primary Tibia: Patients who were implanted with a cemented tibial stem, 5 degree Persona primary tibial component, CCK articular surface, Persona Revision femoral component, and cemented femoral stem.
  Interventions: Device: Persona Revision Knee System
- 8) Primary Splined CCK/CPS/PS with 0 Degree Tibia: Patients with a primary implant (non-revision case) who were implanted with a splined tibial stem, 0 degree Persona Revision tibial component, CCK/PS/CPS articular surface, Persona Revision femoral component, and splined femoral stem.
  Interventions: Device: Persona Revision Knee System
- 9) Primary Cemented CCK/PS/CPS with 0 Degree Tibia: Patients with a primary implant (non-revision case) who were implanted with a cemented tibial stem, 0 degree Persona Revision tibial component, CCK/PS/CPS articular surface, Persona Revision femoral component, and cemented femoral stem.
  Interventions: Device: Persona Revision Knee System
- 10) Primary Cemented CCK/PS/CPS with 5 Degree Primary Tibia: Patients with a primary implant (non-revision case) who were implanted with a cemented tibial stem, 5 degree Persona primary tibial component, CCK/PS/CPS articular surface, Persona Revision femoral component, and cemented femoral stem.
- 11) Infection Cases: Any configuration of PRK components used for end stage (non-temporary) treatment

INTERVENTIONS:
Device: Persona Revision Knee System — Patients in this cohort will have been previously implanted with the Persona Revision Knee system in the described configuration per standard of care. The Persona Revision knee system is a total knee system that is widely available for use in the United States and is designed for use in primary and revision knee surgical interventions.
  Groups: 1) Revision Splined CCK; 2) Revision Cemented CCK; 3) Revision Splined PS/CPS; 4) Revision Cemented PS/CPS; 5) Revision Splined PS/CPS; 6) Revision Cemented PS/CPS; 7) Revision Cemented CCK with 5 Degree Primary Tibia; 8) Primary Splined CCK/CPS/PS with 0 Degree Tibia; 9) Primary Cemented CCK/PS/CPS with 0 Degree Tibia

SUMMARY:
The study will evaluate the performance, clinical benefits and safety of the Persona Revision Knee System in patients who have received primary or revision total knee arthroplasty (TKA) treatment. This will be done using a multicenter, single-arm, consecutive series, retrospective cohort study with prospective follow-up.

DETAILED DESCRIPTION:
Under study are the Persona® Revision Knee System (K181947 and K191625) implants and instrumentation, and any compatible devices being used in conjunction according to the Instructions for Use. This will be accomplished by retrospectively identifying patients who underwent primary or revision TKA with this system and inviting them to participate in prospective data collection at 1, 2, 3, 4, 5, 7, and 10 years postoperative follow-up. As the device was not available for commercial use until late 2019, the retrospective portion will involve those activities that occurred per standard of care for participants.

The primary endpoint for this study will be performance assessed by improvement in the 1989 Knee Society Clinical Rating System (KS) objective knee score (KS-KS) from baseline to 2 years (as evaluated using the overall group mean showing at least the Minimal Clinically Important Difference (MCID) of 5.4 points).

A maximum of 20 sites will contribute to this study. There will be a maximum of 380 patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of at least 18 years of age at the time of screening.
2. Signed an institutional review board approved informed consent.
3. Willingness and ability to comply with the study procedures and visit schedules and ability to understand and follow oral and written post-operative care instructions.
4. Previous medical diagnosis/ history of at least one of the following conditions requiring treatment using the Persona Revision Knee System within a pre-specified study variant configuration (cohort), in accordance with the instructions for use (IFU):

   1. Rheumatoid arthritis, osteoarthritis, traumatic arthritis or polyarthritis
   2. Collagen disorders, and/or avascular necrosis of the femoral condyle
   3. Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy
   4. Moderate valgus, varus, or flexion deformities
   5. The salvage of previously failed surgical attempts or for a knee in which satisfactory stability in flexion cannot be obtained at the time of surgery
5. A pre-operative Knee Society Knee Score (objective assessment) ≤ 80.

Exclusion Criteria:

1) Presence of clinically observed active or suspected latent infection in the affected joint at the time of procedure.

3) Presence of of local/systemic/distant focal infection that may affect or hematogenously spread to the prosthetic joint.

4) Skeletal immaturity or insufficient bone stock on femoral or tibial surfaces which cannot provide adequate support and/or fixation to the prosthesis.

5) Diagnosed with neuropathic arthropathy, osteoporosis, or any loss of musculature or neuromuscular disease that compromises the affected limb.

6) Presence of a stable, painless arthrodesis in a satisfactory functional position in the affected joint.

7) Severe instability of the affected joint secondary to the absence of collateral ligament integrity.

8) Diagnosis of rheumatoid arthritis in conjunction with any of the following at the time of screening:

1. An ulcer of the skin
2. History of recurrent breakdown of the skin
3. Use of steroids

   9) Patient requires simultaneous bilateral knee surgery for treatment of diagnosed condition.

   10) Pregnant or women planning to become pregnant during the time they will be participating in the study.

   11) Any documented clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening which, in the opinion of the Investigator, could compromise patient safety or interfere with the assessment of the safety and treatment effects of the study procedure.

   12) Any patient who is institutionalized, or with a known drug or alcohol dependence currently or within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of a primary or revision total knee procedure who receive Persona Revision Knee implants who meet all the inclusion criteria and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Society Clinical Rating System objective knee score (KS-KS) | 2 years
  The primary endpoint for this study will be performance assessed by improvement in the 1989 Knee Society Clinical Rating System (KS) objective knee score (KS-KS) from baseline to 2 years (as evaluated using the overall group mean showing at least the minimal clinically important difference [MCID] of 5.4 points)
  The Knee Society objective knee score (KS-KS) assesses the knee joint by awarding points for pain, stability, and range of motion, with a minimum possible score of 0 and maximum possible score of 100. As described in Insall et al. (1989), "100 points will be obtained by a well-aligned knee prosthesis with no pain, [at least 121] degrees of motion, and negligible anteroposterior and mediolateral instability."

SECONDARY OUTCOMES:
Incidence and frequency of adverse events. | 2 years
  Safety of the device will be assessed by evaluating the incidence and frequency of adverse events including (re-)revision of any component during the study in accordance with Regulation (EU) 2017/745 - Medical Device Regulation (MDR) Article 80(2) as well as Medical Devices Coordination Group (MDCG) 2020-10/1.
Numeric Rating Scale (NRS) Pain Score | 2 years
  Performance and clinical benefits will be assessed by evaluating improvements in patient reported outcome measures (PROMs) of the Numeric Rating Scale (NRS) pain scores from baseline to 2 years.
  The Numeric Rating Scale (NRS) pain is scored on a scale of 0 to 10. A score of 0 indicates that the patient is experiencing no pain in their knee joint while a score of 10 indicates that the patient is experiencing the worst possible pain in their knee joint.
Knee Injury and Osteoarthritis Outcome Score Junior (KOOS-Jr) | 2 years
  Performance and clinical benefits will be assessed by evaluating improvements in patient reported outcome measures (PROMs) for the Knee Injury and Osteoarthritis Outcome Score Junior (KOOS-Jr) subscale scores from baseline to 2 years.
  The Knee Injury and Osteoarthritis Outcome Score Junior (KOOS-Jr) is scored on a scale of 0 to 100. A score of 100 indicates that a patient is experiencing perfect knee health while a score of 0 indicates that a patient is experiencing total knee disability.

OTHER OUTCOMES:
Radiographic Imaging | 2 years
  Exploratory outcomes will include the evaluation of radiographic imaging as required for adverse event/complication reporting purposes with focus on the following parameters: radiolucency lines, component migration/subsidence, osteolysis, and localized osteopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Jaggard, Study Director — Zimmer Biomet
Locations (16):
- United States (16):
  - Advanced Orthopaedic Specialists, Fayetteville, Arkansas
  - Bowen Hefley Orthopedics, Little Rock, Arkansas
  - Community Foundation Medical Group, Fresno, California
  - Cornerstone Orthopaedics & Sports Medicine, Superior, Colorado
  - Orthopaedic Associates, Inc., Evansville, Indiana
  - Jeff Yergler, LLC, Granger, Indiana
  - Arthroplasty Foundation Inc., Louisville, Kentucky
  - Ascension Providence Rochester Hospital, Rochester, Michigan
  - Michigan Orthopaedic Surgeons, PLLC, Southfield, Michigan
  - TRIA Orthopaedic Center Research Institute, Bloomington, Minnesota
  - Thomas Aleto MD, PC, Columbia, Missouri
  - Orthopaedic Research Institute of New Jersey, Chester, New Jersey
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - ROC Orthopedics, Oregon City, Oregon
  - Penn Medicine/ Lancaster General Health, Lancaster, Pennsylvania
  - Orthopedic Surgeons of Wisconsin, SC, Wauwatosa, Wisconsin